CLINICAL TRIAL: NCT06779292
Title: Application of Multimodal Large Language Models in Emergency Neurology Diagnosis
Brief Title: Application of Large Language Models in Emergency Neurology
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Beijing Institute of Brain Disorders, Capital Medical University, Capital Medical University
Other Study IDs: ALEGN
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Neurology; Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting to the emergency neurology department.
  Interventions: Diagnostic Test: Large Language Model Diagnosis

INTERVENTIONS:
Diagnostic Test: Large Language Model Diagnosis — Using the large language model for diagnosing emergency neurology conditions.

SUMMARY:
Emergency neurology covers a wide range of conditions, often involving urgent situations such as acute cerebrovascular diseases, seizures, central nervous system infections, and consciousness disorders. However, due to the time constraints in emergency care and limited patient information collection, misdiagnosis and missed diagnoses are common issues. Large language models (LLMs) possess powerful natural language processing and knowledge reasoning capabilities, enabling them to directly handle and understand complex, unstructured medical data such as patient medical records, dialogue notes, and laboratory test results. LLMs show broad potential for application in complex medical scenarios. This study aims to evaluate the application value of LLMs in emergency neurology, specifically examining their diagnostic accuracy in emergency neurology conditions, analyzing the feasibility of treatment plans and further examination recommendations proposed by the model, and exploring their potential in improving diagnostic efficiency and aiding decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18-80 years, male or female.
* Patients seeking emergency neurology care.
* Patients who can provide complete medical records (including consultation recordings, physical examination, test results, etc.).
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Patients who directly enter the resuscitation process due to the severity of their condition(e.g., patients who are immediately placed in the ICU).
* Patients with unstable vital signs.
* Patients who are unable to communicate effectively (e.g., severe consciousness impairment or severe cognitive disorders).
* Patients who are currently participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the emergency neurology department
Sampling Method: Probability Sample
Enrollment: 433 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
dignostic accuracy | 1 month
  To evaluate the consistency between the diagnosis made by large language models for emergency patients and the confirmed diagnosis after inpatient or outpatient visits.

SECONDARY OUTCOMES:
Feasibility of treatment plans | 1 month
  Experts use the Emergency Treatment Recommendation Scoring Scale to evaluate the treatment suggestions from conventional methods and large language models. The maximum score is 5 and the minimum score is 1, with 5 representing strong agreement with the recommendation.
dignostic specificity | 1 month
  A comparison of dianostic specificity between large language model diagnosis and emergency department physicians diagnosis
Diagnostic Sensitivity | 1 month
  A comparison of dianostic sensitivity between large language model diagnosis and emergency department physicians diagnosis.
False Discovery Rate | 1 month
  A comparison of the false discovery rate between large language model diagnosis and emergency department physicians diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No